CLINICAL TRIAL: NCT02432703
Title: A Phase 2a Randomized, Double-blind, Placebo-Controlled, Parallel-Group, Multi-center Study Investigating the Efficacy, Safety, and Tolerability of JNJ-42165279 in Subjects With Social Anxiety Disorder.
Brief Title: A Safety and Efficacy Study of JNJ-42165279 in Participants With Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106641; 42165279SAX2001 (Other: Janssen Research & Development, LLC); 2014-004258-32 (EudraCT Number)
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Phobic Disorders
Keywords: Social Anxiety Disorder; JNJ-42165279
MeSH Terms: conditions — Phobic Disorders; Phobia, Social | interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-42165279 (Experimental): Participants will receive 25 milligram (mg) JNJ-42165279 orally once-daily from Day 1 up to 12 weeks.
  Interventions: Drug: JNJ-42165279
- Placebo (Placebo Comparator): Participants will receive a matching placebo orally once-daily from Day 1 up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42165279 — Participants will receive 25 milligram (mg) JNJ-42165279 orally once-daily from Day 1 up to 12 weeks.
  Arms: JNJ-42165279
Drug: Placebo — Participants will receive a matching placebo orally once-daily from Day 1 up to 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy of JNJ-42165279 during 12 weeks of treatment in participants with Social Anxiety Disorder (SAD).

DETAILED DESCRIPTION:
This is a Phase 2a randomized (study drug assigned by chance), double-blind (neither the Investigator nor the participants know about the study intervention), placebo-controlled, parallel-group, multi-center study of JNJ-42165279 in participants with social anxiety disorder. Participants will receive 25 milligram (mg) JNJ-42165279 or matching placebo orally once-daily from Day 1 up to 12 weeks. Participants will primarily be assessed for the change from baseline in Liebowitz Social Anxiety Scale (LSAS) at Week 12. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have a primary DSM-5 diagnosis of Social anxiety disorder (SAD) except those with performance only as a specifier. Participants with a diagnosis of comorbid Generalized Anxiety Disorder (GAD) or Major Depressive Disorder (MDD) may be included if the Investigator considers SAD to be the predominant diagnosis. Participants with current or lifetime history of Attention deficit hyperactivity disorder (ADHD) and specific phobia may be included as well
* Must have a Liebowitz Social Anxiety Scale score greater than or equal (>=) 70 at Screening and Baseline
* Participants with a current episode of MDD must have a HDRS17 total score less than or equal to (<=) 18
* Must have a body mass index (BMI) between 18 and 35 kilogram per meter square (kg/m^2), inclusive, at screening
* Female participants must be either postmenopausal or surgically sterile

Exclusion Criteria:

* Participants who have performance only SAD are excluded. Participants with other current significant psychiatric condition(s) (Axis 1 under DSM-IV), including, but not limited to, MDD with psychotic features (lifetime), bipolar disorder (including lifetime diagnosis), obsessive-compulsive disorder, borderline personality disorder, eating disorder (e.g., bulimia, anorexia nervosa), autism spectrum disorders, post-traumatic stress disorder (PTSD) or schizophrenia are excluded. Participants with a diagnosis of comorbid GAD or MDD may be included
* Participants is currently receiving specific psychotherapy for SAD
* Has a history of more than two unsuccessful adequate pharmacological treatment trials for SAD, defined as lack of response to at least 10 weeks of treatment at adequate doses (e.g., paroxetine >= 40 milligram per day (mg/day) or its equivalent; or clonazepam >= 2.5 mg/day or its equivalent)
* Concurrent use of psychotropic medications
* has a history of or current thyroid disease, thyroid dysfunction and is currently untreated for it

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- United States (13):
  - La Jolla, California
  - Hartford, Connecticut
  - Orlando, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Natick, Massachusetts
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Allentown, Pennsylvania
  - Reading, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
- Australia (4):
  - Adelaide
  - Frankston
  - Melbourne
  - Perth
- Canada (4):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Mississauga, Ontario
  - Toronto, Ontario

REFERENCES:
- [Derived] Schmidt ME, Liebowitz MR, Stein MB, Grunfeld J, Van Hove I, Simmons WK, Van Der Ark P, Palmer JA, Saad ZS, Pemberton DJ, Van Nueten L, Drevets WC. The effects of inhibition of fatty acid amide hydrolase (FAAH) by JNJ-42165279 in social anxiety disorder: a double-blind, randomized, placebo-controlled proof-of-concept study. Neuropsychopharmacology. 2021 Apr;46(5):1004-1010. doi: 10.1038/s41386-020-00888-1. Epub 2020 Oct 18. PMID 33070154

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among 150 participants, one participant was randomized by error. Only 149 participants received treatment and were included in the analysis.
Groups:
- Placebo: Participants with social anxiety disorder (SAD) received matching placebo orally once daily for 12 weeks.
- JNJ-42165279 25 mg: Participants with SAD received JNJ-42165279 25 milligrams (mg) orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | JNJ-42165279 25 mg
Started | 75 | 74
Completed | 53 | 56
Not Completed | 22 | 18
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Other | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-42165279 25 mg | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (13.65) | 38.3 (12.53) | 37.8 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 49 | 48 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 22
  Not Hispanic or Latino | 66 | 61 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 45 | 50 | 95
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 11 | 12 | 23
  CANADA | 14 | 12 | 26
  UNITED STATES | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Liebowitz Social Anxiety Scale (LSAS) Total Score
Description: The LSAS is a 24-item, semi-structured interview on the severity of Social Anxiety Disorder. The LSAS separately assesses fear and avoidance of 24 social situations. The scale is divided into 2 subscales, 13 situations concerning performance anxiety, and 11 situations pertaining to social situations. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations (0=none, 1=mild, 2=moderate, 3= severe), and then the same items are rated regarding avoidance of the situation (0=never, 1=occasionally, 2=often, 3=usually) with higher scores indicating greater social anxiety. The LSAS fear/anxiety and avoidance subscale was calculated by summing the 24 fear/anxiety and avoidance item scores of the LSAS, and ranges from 0 to 72. Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points and a minimum of 0 points. Higher scores indicated higher probability of social anxiety disorder (SAD).
Time Frame: Baseline and Week 12
Population: Intent-to-treat (ITT) analysis set included all randomized participants who received at least 1 dose of the study agent (either placebo or JNJ-42165279), and had at least 1 assessment in the double-blind treatment phase on any of the efficacy parameters.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale | -22.4 (23.57) | -29.4 (27.47)

2. Secondary Outcome: Change From Baseline in LSAS Fear/Anxiety and Avoidance Subscales
Description: The LSAS is a 24-item, semi-structured interview on the severity of Social Anxiety Disorder. The LSAS separately assesses fear and avoidance of 24 social situations. The scale is divided into 2 subscales, 13 situations concerning performance anxiety, and 11 situations pertaining to social situations. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations (0=none, 1=mild, 2=moderate, 3= severe), and then the same items are rated regarding avoidance of the situation (0=never, 1=occasionally, 2=often, 3=usually). Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points and a minimum of 0 points. Higher scores indicated higher probability of SAD. The LSAS fear/anxiety and avoidance subscale was calculated by summing the 24 fear/anxiety and avoidance item scores of the LSAS, and ranges from 0 to 72.
Time Frame: Baseline and Week 12
Population: ITT analysis set included all randomized participants who received at least 1 dose of the study agent (either placebo or JNJ-42165279), and had at least 1 assessment in the double-blind treatment phase on any of the efficacy parameters.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale
  Fear/Anxiety | -10.7 (12.31) | -14.6 (13.65)
  Avoidance | -11.7 (12.16) | -14.9 (14.45)

3. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 50 Percent (%) Improvement From Baseline (Responders) on LSAS Total Score
Description: Responders are participants with >= 50% improvement from baseline. The LSAS scale consists of 24 items which are divided into 2 subscales that address social interactional (11 items) and performance (13 items) situations. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations (0=none, 1=mild, 2=moderate, 3= severe), and then the same items are rated regarding avoidance of the situation (0=never, 1=occasionally, 2=often, 3=usually) with higher scores indicating greater social anxiety. The LSAS fear and avoidance subscale was calculated by summing the 24 fear/anxiety and avoidance item scores of the LSAS, and ranges from 0 to 72. Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points and a minimum of 0 points. Higher scores indicated higher probability of SAD.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
percentage of participants | 12.7 | 18.6

4. Secondary Outcome: Percentage of Participants With >=30% Improvement From Baseline (Remitters) on LSAS Total Score
Description: Remitters are participants with >= 30% improvement from baseline on LSAS total score. The LSAS scale consists of 24 items which are divided into 2 subscales that address social interactional (11 items) and performance (13 items) situations. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations (0=none, 1=mild, 2=moderate, 3= severe), and then the same items are rated regarding avoidance of the situation (0=never, 1=occasionally, 2=often, 3=usually) with higher scores indicating greater social anxiety. The LSAS fear and avoidance subscale was calculated by summing the 24 fear/anxiety and avoidance item scores of the LSAS, and ranges from 0 to 72. Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points and a minimum of 0 points. Higher scores indicated higher probability of SAD.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
percentage of participants | 23.6 | 42.4

5. Secondary Outcome: Change From Baseline in Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A) Total Score
Description: The SIGH-A was included to determine the frequency and severity of signs and symptoms of anxiety, including participants with comorbid generalized anxiety disorders (GAD) and major depressive disorder (MDD), and determine both their influence on treatment and their responsiveness to treatment. The SIGH-A scale consists of 14 items with a score of 0 to 4. Higher scores indicated higher severity (0-absent, 1-mild, 2-moderate, 3-severe, 4-incapacitating). The SIGH-A total score was calculated by summing the 14 item scores, and ranges from 0 to 56. Higher scores indicated worse results.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale | -3.0 (6.20) | -4.2 (5.90)

6. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM)-A6 Score
Description: The HAM-A6 is a 6-item subscale derived from the original Hamilton Anxiety scale (HAM-A). It comprises of five psychic anxiety symptoms: anxious mood, psychic tension, fears, intellectual disturbances, and anxious behavior observed at the interview, as well as one somatic item, muscular tension. Each of the 6 items is rated by the clinician on a 5-point scale ranging from 0 (not present) to 4 (maximum degree). The HAM-A6 score was calculated by summing the 6 item scores, and ranges from 0 to 24. Higher scores indicated greater severity of symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale | -1.9 (3.32) | -2.3 (3.79)

7. Secondary Outcome: Change From Baseline in Hamilton Depression Rating Scale (HDRS)-17 Total Score
Description: The HDRS-17 is a clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale | -0.9 (4.71) | -1.8 (3.99)

8. Secondary Outcome: Change From Baseline in HDRS17 Anxiety/Somatization Factor Total Score
Description: The HDRS17 anxiety/somatization factor derived from Cleary and Guy's factor analysis of the HDRS17 scale, includes six items from the original 17-item version: the items for psychic anxiety, somatic anxiety, gastrointestinal somatic symptoms, general somatic symptoms, hypochondriasis, and insight. Each of these items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). HDRS17 anxiety/somatization factor total score was calculated as the sum of the 6 item scores ranging from 0 to 18. Higher scores indicated greater severity of symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale | -0.4 (2.25) | -0.9 (2.05)

9. Secondary Outcome: Change From Baseline in HAM-D6 Total Score
Description: A 6-item subscale from the HDRS17 (HAM-D6) was analyzed as it had been shown to be a uni-dimensional scale that provided information to core depressive symptoms and was sensitive to treatment response. The six items were: depressed mood, guilt feelings, work and interests, psychomotor retardation, psychic anxiety, and general somatics (tiredness and pains). Each of these items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). General somatics is scored 0 to 2 and all others are scored 0 to 4. The HAM-D6 total score was calculated by summing the 6 items scores, and ranges from 0 to 22. Higher scores indicated greater severity of core symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
units on a scale | -0.7 (2.89) | -1.0 (2.56)

10. Secondary Outcome: Percentage of Participants With Change From Baseline in Clinical Global Impression- Improvement (CGI-I) Score
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention. The CGI-I is rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Percentage of participants with change from baseline (very much improved or much improved and Worsening or no change) in CGI-I score were reported.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of the study agent (either placebo or JNJ-42165279), and had at least 1 assessment in the double-blind treatment phase on any of the efficacy parameters.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
percentage of participants
  Very much improved or much improved | 23.6 | 44.1
  Worsening or no change | 45.5 | 35.6

11. Secondary Outcome: Percentage of Participants With >=50% Improvement From Baseline (Responders) in SIGH-A Total Score
Description: Responders are participants with >= 50% improvement from baseline in SIGH-A total score. The SIGH-A scale consists of 14 items with a score of 0 to 4. Higher scores indicated higher severity (0-absent, 1-mild, 2-moderate, 3 severe, 4-incapacitating). The SIGH-A total score was calculated by summing the 14 item scores, and ranges from 0 to 56. Higher scores indicated worse results.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42165279 25 mg
Number analyzed (Participants) | 68 | 66
percentage of participants | 47.3 | 45.6

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: Safety analysis set included all randomized participants who received at least one dose of study medication (either placebo or JNJ-42165279).
Arm/Group | Placebo | JNJ-42165279 25 mg
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 2/74
Other Adverse Events (participants affected / at risk) | 27/75 | 26/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | JNJ-42165279 25 mg (N=74)
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Alcohol Use Disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | JNJ-42165279 25 mg (N=74)
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 3 | 6
Nasopharyngitis (Infections and infestations) | 6 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 5
Headache (Nervous system disorders) | 13 | 15
Insomnia (Psychiatric disorders) | 6 | 1

LIMITATIONS AND CAVEATS:
The US food and drug administration placed a clinical hold on studies being conducted with fatty acid amide hydrolase (FAAH) inhibitor. When determined that serious adverse events were not related to FAAH inhibition, Janssen resumed this study in December 2016. At time of study suspension, an unblinded safety analysis was performed, and hence sample size was increased to replace participants who withdrew due to study suspension. Planned analyses were performed at time of final database lock.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02432703/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT02432703/SAP_001.pdf